CLINICAL TRIAL: NCT06319365
Title: The Effect of Yoga on Hypertensive Women's Blood Pressure, Sexual Life, And Marital Compliance:Randomized Controlled Trial
Brief Title: Yoga on Women's Blood Pressure, Sexual Life, And Marital Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Gürcan Solmaz, Principal investigator, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: gurcansolmaz
Record Dates: First submitted 2024-03-10; First posted 2024-03-20 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Hypertension; Sexuality
Keywords: yoga, hypertension, sexality, women
MeSH Terms: conditions — Hypertension; Sexuality | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- yoga group (Experimental): the yoga practice of the group should be completed at the end of 12 weeks. Participants should be encouraged to practice at home 3 days a week for 3 months. An example of yoga practices in the research for women should be shared as a video.
  Interventions: Behavioral: yoga
- control group (No Intervention): The control group should be continue standard hypertension treatment

INTERVENTIONS:
Behavioral: yoga — the yoga practice of the group should completed at the end of 12 weeks
  Arms: yoga group

SUMMARY:
Introduction This study will examine the effects of a 12-week yoga program consisting of one-hour sessions three times a week on blood pressure, sexual life and marital adjustment among hypertensive women. Hypertension can adversely affect vascular health and affect marital relationships by contributing to sexual dysfunction.

Method. The study will be a pre-post test randomized controlled study in accordance with CONSORT rules. Personal Information Form, Bloood pressure measurement, Arizona Sexual Experience Scale and Marital Adjustment Test will be used for data collection.

DETAILED DESCRIPTION:
Factors such as hormonal changes, oral contraceptive use, obesity, and stress level increase hypertension (HT) predisposition in women. Despite the use of many antihypertensive drugs, less than a third of women undergoing treatment can achieve the targeted blood pressure. Therefore, different strategic approaches are needed to reduce blood pressure. Wolff (2016) shows that yoga provides a decrease in systolic blood pressure (SBP) by up to 6 mmHg and diastolic blood pressure (DBP) by up to 5 mmHg, 12-week yoga study conducted with a home video for women showed that DBP decreased according to the first measurements, it has been determined that the quality of life has increased. High blood pressure that cannot be controlled can cause deterioration in sexual functions as well as damage to many organs. Since HT produces negative effects on the vascular system, sexual dysfunctions may occur. Although the number of studies on the relationship between HT and sexual functions is limited, the issue has been discussed especially in terms of the sexual life of men These vascular changes can cause sexual reluctance in women by negatively affecting the clitoral and vaginal vascular structure, decreased blood flow in the pelvic region, thinning of the vaginal wall smooth muscles, vaginal dryness, and pain during sexual intercourse, orgasm, and arousal phase. In one of the few studies, it was determined that 42% of hypertensive women experience sexual dysfunction. The sexual life of women may be adversely affected as a result of the menopause process, the side effects of antihypertensive treatment, and the physiological changes induced by HT in the body. Marriage is one of the areas in which the quality of life plays the most active role. Sexual life, which is negatively affected, can harm marital compliance over time. Marital problems can negatively affect women's blood pressure. At this point, there is a need for programs that will help women maintain both their physical and psychological health. Yoga is a practice that provides physical and mental flexibility without side effects in maintaining and improving health. In the studies on yoga, it has been determined that body awareness is higher in people who do yoga and that doing yoga reduces anxiety. When studies on the changes in women who practice yoga are examined; significant improvement was found in issues such as stress, depression, body image, incontinence, and sexuality. In a study, yoga program applied to women with incontinence problems, it reduced the inflammatory process associated with incontinence because most of the yoga asanas stretch the pelvic floor muscles ,and could be applied as a complementary treatment. Asanas such as Mula Bandha (Root lock) stretch the pelvic floor muscles, accelerate blood flow in the genital area and have similar effects to kegel exercises and provide improvement in sexual desire, arousal, vaginal hydration, orgasm, pain and sexual satisfaction. Considering the positive effects of yoga on blood pressure and sexual life, it can be interpreted that it may have positive reflections on marriage. No study was found that evaluated the solutions for the blood pressure and sexual life problems experienced by married hypertensive women. It is the first in terms of study subject and design.

Method. The study will be a pre-post test randomized controlled study in accordance with CONSORT rules. Personal Information Form, Bloood pressure measurement, Arizona Sexual Experience Scale and Marital Adjustment Test will be used for data collection.

ELIGIBILITY:
Inclusion Criteria:

* (a) women aged 18 years or older; (b) Those who have been diagnosed with hypertension for at least three months and whose treatment continues; (c) Those who are not pregnant; (d) are married; (e) Those who have the equipment (computer, smartphone or tablet) to participate in the yoga program online (f) Those who want to participate in the research.

Exclusion Criteria:

* a) the illiterate; (b) Those who do not want to participate in the research; (c) Having a severe mental disorder; (e) Those who, with the opinion of an expert, had any condition that would hinder the practice of yoga were not included in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 70 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
blood presure | 3 months
  sistolic blood presure and diastolic blood pressure mensurement

CONTACTS AND LOCATIONS:
Overall Officials: Gürcan Solmaz, PhD, Study Director — İstanbulUniversity-Cerrahpaşa
Locations (1):
- Yalova University, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No